CLINICAL TRIAL: NCT04358601
Title: Migration and Survival of All-polyethylene Tibial Components Compared to the Metal-backed Modular Components of the Triathlon PS Total Knee System. A RSA Study
Brief Title: All-poly Versus Metal-backed
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Allpoly Triathlon PS
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All-polyethylene tibial components (Experimental): Triathlon PS Knee System with all-polyethylene tibial components
  Interventions: Device: Triathlon PS Knee System with all-polyethylene tibial components
- Metal-backed modular components (Active Comparator): Triathlon PS Knee System with metal-backed modular components
  Interventions: Device: Triathlon PS Knee System with metal-backed modular components

INTERVENTIONS:
Device: Triathlon PS Knee System with all-polyethylene tibial components — Primary Total Knee Replacement
  Other Names: Stryker Orthopaedics
  Arms: All-polyethylene tibial components
Device: Triathlon PS Knee System with metal-backed modular components — Primary Total Knee Replacement
  Other Names: Stryker Orthopaedics
  Arms: Metal-backed modular components

SUMMARY:
The primary objective is the assessment of prosthetic migration results after two years of the Triathlon PS Knee System with all-polyethylene tibial components compared to the Triathlon PS Knee System with metal-backed modular components by means of Roentgen Stereophotogrammetry.

DETAILED DESCRIPTION:
The secondary objective will be the prediction of the long-term survival based on the two-year migration patterns combined with clinical factors and radiographic aspects. In order to identify other clinical parameters besides the fixation of the prosthesis components, clinical scores and radiographic aspects will be correlated with the RSA outcome.

ELIGIBILITY:
1. The subject is morbidly obese, defined as Body Mass Index (BMI) of > 40. 2. Patient has a flexion contracture of 15° and more. 3. Patient has a varus/valgus contracture of 15° and more. 4. Patients with a pre-operative knee score of >70. 5. The subject has a history of total or unicompartmental reconstruction of the affected joint. 6. The subject will be operated bilaterally. 7. Patients who had a Total Hip Arthroplasty (THA) on contralateral and/or ipsilateral side within the last year that is considered to have an unsatisfactory outcome (Patients with contralateral and/or ipsilateral THA > 1 year ago with good outcome can be included in the study). 8. Patients who had a Total Knee Arthroplasty (TKA) on contralateral side within the last 6 months that is considered to have an unsatisfactory outcome. (Patients with contralateral TKA > 6 months ago with good outcome can be included in the study). 9. The subject has an active or suspected latent infection in or about the knee joint. 10. Osteomyelitis 11. Sepsis 12. Patient who is expected to need lower limb joint replacement for another joint within one year. 13. The subject has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device. 14. The subject has a systemic or metabolic disorder leading to progressive bone deterioration. 15. The subject is immunologically suppressed or receiving steroids in excess of normal physiological requirements. 16. The subject's bone stock in compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis. 17. The subject has had a knee fusion to the affected joint. 18. Female patients planning a pregnancy during the course of the study. 19. The patient is unable or unwilling to sign the Informed Consent specific to this study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Migration, measured by means of RSA | 2 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA)

SECONDARY OUTCOMES:
Migration, measured by means of RSA | 10 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA)
Investigation of clinical performance and patient outcome with the Knee Society Score (KSS) | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Investigation of clinical performance and patient outcome with the Knee Injury and Osteoarthritis Outcome Score (KOOS) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  KOOS consists of 5 subscales: Pain, other symptoms, function in daily living , function in sport and recreation and knee related quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms).
Investigation of clinical performance and patient outcome with EuroQuol-5 dimension (EQ-5D) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
Investigation of clinical performance and patient outcome with the Forgotten Joint Score (FJS) patient questionnaire. | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The FJS consists of 12 questions and focuses on the patients' awareness of their joint replacement during a range of day to day and recreational activities. The score has a range of 0-100.questionnaire
Investigation of patient outcome with radiographic analysis | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  Plain radiographs will be obtained for assessment of fixation of the device.